CLINICAL TRIAL: NCT04584086
Title: Changes in the MRI Signal in Patients With Benign Tumors of the Brain and Meninges Treated With Proton Therapy: Impact of TEL and the Biological Dose Received
Acronym: BRAIN TEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A02023-36
Record Dates: First submitted 2020-10-01; First posted 2020-10-12 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Benign Brain Tumors; Proton Therapy
Keywords: MRI
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI 3 Tesla (Experimental): Patients will be followed by 3 Tesla MRIs during the study
  Interventions: Device: MRI 3 tesla

INTERVENTIONS:
Device: MRI 3 tesla — 1.5 Tesla MRIs, usually used as pre-treatment and, between 3 and 6 months after irradiation, are replaced in the study by 3 Tesla MRIs (pre-treatment and at 6 months)
  In addition, two additional MRIs, also performed with a 3 Tesla magnetic field, will be performed:
  * During treatment when half of the prescribed dose has been delivered.
  * 1 month after the end of the irradiation.

SUMMARY:
The main objective is to detect with TESLA multiparametric 3 MRI, the MRI secondary changes to protontherapy irradiation and to correlate them with TEL mapping, physical dose and biological dose. A model should thus be able to be proposed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven or highly probable grade I meningiomas, histologically proven grade II meningiomas.
* Only meningiomas of the anterior and middle floors of the base of the skull are included.
* Indication of proton therapy retained in RCP and / or proton therapy technical staff (Caen site)
* Patient aged 18 or over
* Patient affiliated to a social security scheme
* Signature of informed consent before any specific procedure related to the study

Exclusion Criteria:

* History of brain or face irradiation.
* Implant or foreign body that can alter MRI imaging.
* Contraindication to MRI (pace maker, claustrophobia ...) - Hypersensitivity to gadoteric acid, to meglumine or to any medicine containing gadolinium
* Genetic radio sensitizing syndrome
* Known neurological comorbidities (stroke, Parkinson's, etc.) that may impact MRI data.
* Simultaneous participation in a therapeutic clinical trial
* Patient unable to undergo the trial follow-up for geographic, social or psychopathological reasons
* Pregnant or breastfeeding women
* Persons deprived of their liberty (see article L 1121-6 CSP),
* Adults who are the subject of a legal protection measure or unable to express their consent (see article L 1121-8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluate by TESLA multiparametric 3 MRI the modifications of the MRI signal :Change from Baseline at 1, 3 and 6 months | Up to 6 months
  modifications of the MRI signal on the various sequences carried out, during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No